CLINICAL TRIAL: NCT06768645
Title: The Effectiveness of Diabetic Foot Wound Prevention Training Given With Pecha Kucha (20*20) Presentation Technique: A Randomized Controlled
Brief Title: The Effectiveness of Diabetic Foot Wound Prevention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Nursing Associate Professor, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulMU
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Patient Education; Diabetic Foot Ulcer; PechaKucha Method
Keywords: Pecha Kucha; Type 2 diabetes; Diabetic Foot; Patient Education
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Assuming a power of 80% and an α risk of. 05, a sample size of 120 was determined to be appropriate. Considering the possibility of missing data, the study initially included 65 participants in both the experimental and control groups. A computer-based random number generator was used for group assignment, and allocation concealment was ensured by using sealed envelopes containing random numbers opened by a separate researcher. The study was completed with 62 participants in the experimental group and 63 in the control group, due to some participants withdrawing.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecha Kucha (Experimental): Given Pecha Kucha education
  Interventions: Behavioral: Diabetic foot care education delivered using the Pecha Kucha method
- Control (Active Comparator): normal education
  Interventions: Behavioral: traditional diabetic foot care education

INTERVENTIONS:
Behavioral: Diabetic foot care education delivered using the Pecha Kucha method — The study commenced after obtaining ethical approval and written consent from the relevant institution. The Pecha Kucha presentation was prepared by the researcher, adhering to established literature and the specific requirements of the technique. The education covered six key topics: 1) Diabetes and Foot Problems, 2) Daily Foot Care, 3) Appropriate Socks, 4) Appropriate Footwear, 5) Nail Care, and 6) Daily Life Precautions. Expert opinions were sought from four academics (S.Ö; K.L; Z.Z; G.F) with expertise in the field to establish content validity for the final version of the Pecha Kucha diabetic foot care presentation. Following expert approval, a pilot study was conducted with 10 diabetic patients who met the sample group criteria. Feedback from these patients regarding system functionality, clarity, and flow was incorporated to finalize the presentation. Afterward, the finalized "Pecha Kucha Information" training was delivered to the experimental group. The presentations were cond
  Arms: Pecha Kucha
Behavioral: traditional diabetic foot care education — traditional diabetic foot care education
  Arms: Control

SUMMARY:
This study aimed to evaluate the impact of diabetic foot care training delivered using the Pecha Kucha (20*20) presentation method on the knowledge, self-efficacy, and behavior levels of patients with Type 2 diabetes. Conducted between December 10, 2023, and October 7, 2024, this randomized controlled experimental study included 125 diabetic individuals, with 62 in the experimental group and 63 in the control group. The experimental group received diabetic foot care education using the Pecha Kucha method, while the control group received conventional education. Data were collected using the Patient Assessment Form, Diabetes Foot Knowledge Questionnaire, Diabetic Foot Care Self-Efficacy Scale, and Foot Self-Care Behavior Scale.

DETAILED DESCRIPTION:
This study aimed to evaluate the impact of diabetic foot care training delivered using the Pecha Kucha (20*20) presentation method on the knowledge, self-efficacy, and behavior levels of patients with Type 2 diabetes. Conducted between December 10, 2023, and October 7, 2024, this randomized controlled experimental study included 125 diabetic individuals, with 62 in the experimental group and 63 in the control group. The experimental group received diabetic foot care education using the Pecha Kucha method, while the control group received conventional education. Data were collected using the Patient Assessment Form, Diabetes Foot Knowledge Questionnaire, Diabetic Foot Care Self-Efficacy Scale, and Foot Self-Care Behavior Scale.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes according to the American Diabetes Association (ADA) criteria at least six months before the study
* age 18 years or older, literacy in and ability to speak Turkish,
* absence of communication/mental problems,
* willingness to participate in the study.

Exclusion Criteria:

* presence of advanced retinopathy, violation of inclusion criteria, withdrawal of consent by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Diabetes Foot Knowledge Questionnaire | up to 24 weeks
  Diabetes Foot Knowledge Questionnaire min:0 max: 5 , Above average placement
Diabetic Foot Care Self-Efficacy Scale | up to 24 weeks
  Diabetic Foot Care Self-Efficacy Scale min:0 max:100 , scores above the 50 points
Foot Self-Care Behavior Scale | up to 24 weeks
  Foot Self-Care Behavior Scale min: 10 max :86, scores above the 48 point

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dincer B, Kocali C, Elveren T, Demir S, Demir K, Dolu FN, Feyizoglu G. The Effectiveness of Diabetic Foot Wound Prevention Training Given with Pecha Kucha (20*20) Presentation Technique: A Randomized Controlled. Int J Low Extrem Wounds. 2025 Feb 13:15347346251318778. doi: 10.1177/15347346251318778. Online ahead of print. PMID 39943850